CLINICAL TRIAL: NCT02815709
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo and Active-controlled Study of Oliceridine (TRV130) for the Treatment of Moderate to Severe Acute Pain After Bunionectomy
Brief Title: Study of Oliceridine (TRV130) for the Treatment of Moderate to Severe Acute Pain After Bunionectomy
Acronym: APOLLO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP130-3001
Record Dates: First submitted 2016-05-12; First posted 2016-06-28 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Treatment 1 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Treatment 2 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Treatment 3 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Morphine (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Oliceridine
  Arms: Treatment 1 Oliceridine; Treatment 2 Oliceridine; Treatment 3 Oliceridine
Drug: Placebo
  Arms: Placebo
Drug: Morphine
  Arms: Morphine

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of intravenous (IV) oliceridine administered as needed (PRN) compared with placebo in patients with moderate to severe acute postoperative pain after bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone primary, unilateral, first metatarsal bunionectomy (osteotomy and internal fixation) with no additional collateral procedures.
* Experiences a pain intensity rating of moderate to severe acute pain.
* Able to provide written informed consent before any study procedure.

Exclusion Criteria:

* ASA Physical Status Classification System classification of P3 or worse.
* Has surgical or post-surgical complications.
* Has clinically significant medical conditions or history of such conditions that may interfere with the interpretation of efficacy, safety, or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Has previously participated in another TRV130 clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, MD, Study Director — Trevena Inc.
Locations (7):
- United States (7):
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Pasadena, California
  - Research Site, Pasadena, Maryland
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Resarch Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-Surgical Entry Criteria
Groups:
- Treatment 1 Oliceridine: Oliceridine 0.1 mg
- Treatment 2 Oliceridine: Oliceridine 0.35 mg
- Treatment 3 Oliceridine: Oliceridine 0.5 mg
- Placebo: Placebo
- Morphine: Morphine
Period: Overall Study
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
Started | 82 | 86 | 82 | 84 | 84
Treated With Study Medication | 76 | 79 | 79 | 79 | 76
Completed | 75 (Completed Study) | 78 (Completed Study) | 75 (Completed Study) | 76 (Completed Study) | 74 (Completed Study)
Not Completed | 7 | 8 | 7 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine | Total
Number analyzed (Participants) | 76 | 79 | 79 | 79 | 76 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 73 | 75 | 76 | 70 | 363
  >=65 years | 7 | 6 | 4 | 3 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.65) | 43.6 (13.91) | 46.9 (13.81) | 44.1 (12.58) | 43.3 (14.13) | 45.1 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 66 | 70 | 65 | 330
  Male | 12 | 14 | 13 | 9 | 11 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 25 | 19 | 17 | 18 | 96
  Not Hispanic or Latino | 59 | 54 | 60 | 62 | 58 | 293
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 47 | 56 | 61 | 56 | 50 | 270
  Black or African American | 22 | 17 | 13 | 21 | 21 | 94
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 1 | 4
  Asian | 4 | 4 | 1 | 1 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 0 | 0 | 4
  Other | 1 | 1 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 76 | 79 | 79 | 79 | 76 | 389

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Respond to Study Medication at the 48-hr Numeric Pain Rating Scale (NRS) Assessment Compared to Placebo.
Time Frame: 48 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
Number analyzed (Participants) | 76 | 79 | 79 | 79 | 76
Participants | 38 | 49 | 52 | 12 | 54

2. Secondary Outcome: Number of Respiratory Safety Events Compared to Morphine.
Time Frame: 48 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Number; unit: Respiratory Safety Events
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
Number analyzed (Participants) | 76 | 79 | 79 | 79 | 76
Respiratory Safety Events | 1 | 7 | 11 | 0 | 14

3. Secondary Outcome: Duration of Respiratory Safety Events Compared to Morphine.
Time Frame: 48 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Mean (Standard Error); unit: hours
Groups:
- Treatment 2 Oliceridine: Oliceridine 0.35
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
Number analyzed (Participants) | 76 | 79 | 79 | 79 | 76
hours | 2.21 (1.796) | 3.44 (1.186) | 3.34 (0.797) | 2.94 (1.074) | 5.14 (1.060)

4. Secondary Outcome: Odds Ratio of Patients Who Respond to Study Medication at the 48-hr NRS Assessment Compared to Morphine.
Description: Odds ratio of 48-hour responder analysis versus morphine. Number of patients who responded to study medication at the 48-hr NRS assessment is captured in the primary outcome measure.
Time Frame: 48 hours
Population: The analysis population reflects the number of patients treated with study medication. The morphine and placebo Arms/Groups are not included, as this is a comparison of study medication against morphine.
Measure: Number; unit: odds ratio
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine
Number analyzed (Participants) | 76 | 79 | 79
odds ratio | 1.5 | 2.54 | 2.89

5. Secondary Outcome: Number of Patients With Treatment-related Adverse Events.
Time Frame: 48 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
Number analyzed (Participants) | 76 | 79 | 79 | 79 | 76
Participants | 48 | 59 | 65 | 32 | 68

ADVERSE EVENTS:
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Placebo | Morphine
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/79 | 0/79 | 0/79 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/79 | 0/79 | 0/79 | 0/76
Other Adverse Events (participants affected / at risk) | 56/76 | 68/79 | 72/79 | 54/79 | 73/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 Oliceridine (N=76) | Treatment 2 Oliceridine (N=79) | Treatment 3 Oliceridine (N=79) | Placebo (N=79) | Morphine (N=76)
Nausea (Gastrointestinal disorders) | 27 | 44 | 50 | 19 | 49
Vomiting (Gastrointestinal disorders) | 13 | 31 | 32 | 5 | 38
Dizziness (Nervous system disorders) | 21 | 25 | 28 | 8 | 26
Headache (Nervous system disorders) | 19 | 20 | 26 | 24 | 23
Somnolence (Nervous system disorders) | 4 | 15 | 10 | 5 | 10
Constipation (Gastrointestinal disorders) | 8 | 9 | 11 | 9 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 12 | 3 | 6 | 15
Hot Flush (Vascular disorders) | 2 | 3 | 6 | 1 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7 | 0 | 7
Dry Mouth (Gastrointestinal disorders) | 1 | 4 | 4 | 1 | 12
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 2 | 3
Sedation (Nervous system disorders) | 2 | 4 | 3 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 4 | 3 | 1 | 3
Oxygen Saturation Decreased (Investigations) | 1 | 3 | 4 | 0 | 7
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 4 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 9
Infusion Site Extravasation (General disorders) | 2 | 0 | 3 | 6 | 2
Chest Discomfort (General disorders) | 0 | 1 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other